CLINICAL TRIAL: NCT05957328
Title: Effect of Ferrous Ascorbate Versus Liposomal Iron on Hemoglobin Concentration and Iron Indices in 6 to 59 Months Age Children With Nutritional Iron-Deficiency Anemia: A Double-blinded Single Centre Randomized Clinical Trial
Brief Title: A Study to Compare Liposomal Iron With Ferrous Ascorbate in the Treatment of Iron Deficiency Anemia in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Namita Mishra, Associate Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AIIMS/RBL/IRC/69/2022
Record Dates: First submitted 2023-06-01; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Nutritional Anemia
Keywords: iron deficiency anemia; liposomal iron; under 5 children
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- liposomal iron group (Active Comparator): The group would be given liposomal iron syrup at a dose of 1mg per kg per day once a day for 3 months
  Interventions: Drug: Ferric Pyrophosphate Liposomal
- ferrous ascorbate group (Active Comparator): The group would be given ferrous ascorbate syrup at a dose of 3mg per kg per day once a day for 3 months
  Interventions: Drug: ferrous ascorbate

INTERVENTIONS:
Drug: Ferric Pyrophosphate Liposomal — Liposomal iron, a form of ferric pyrophosphate is transported within a phospholipid membrane, absorbed by the intestinal M cells, reaches to the liver directly through lymphatics and finally released. Due to this mechanism, liposomal iron has been reported to have better bioavailability than traditional iron preparations thus requiring lesser dose and producing fewer adverse effects The group would be given liposomal iron syrup at a dose of 1mg per kg per day once a day for 3 months
  Other Names: liposomal iron
  Arms: liposomal iron group
Drug: ferrous ascorbate — one of the most commonly used forms of iron syrup in children. The group would be given ferrous ascorbate syrup at a dose of 3mg per kg per day once a day for 3 months
  Other Names: Feronia XT,
  Arms: ferrous ascorbate group

SUMMARY:
This trial is designed to compare the efficacy of ferrous ascorbate versus liposomal iron for the treatment of nutritional iron deficiency anemia (IDA) amongst 6 to 59 months age children as determined by the increase in hemoglobin concentration and change in iron indices after 12 weeks of treatment. This study will be a randomized double-blinded single-center study done at the outpatient department of the Department of Pediatrics. All the children between 6 months to 59 months with nutritional IDA will be enrolled in the study. Written informed consent will be taken from the caregiver. At baseline detailed history will be taken and a complete physical examination will be done. Complete blood count (CBC), Peripheral smear, corrected reticulocyte count, Serum iron, Serum ferritin, and serum Total iron binding capacity(TIBC) will be done at baseline. Transferrin saturation will be calculated with the formula Serum Iron/ TIBC ×100. C Reactive Protein (CRP) and alpha1- acid glycoprotein (AGP) will be done to look for inflammation. Eligible subjects would be randomized in a 1:1 ratio by computerized software to receive either ferrous ascorbate or liposomal iron. Subjects in the ferrous ascorbate group would be given the drug at a dose of 3mg/kg/day OD of elemental iron. Subjects in the liposomal group would be given 1mg/kg/day OD of liposomal iron. Follow-up visits would be done at 4 and 12 weeks. Follow-up at 4 weeks is required to check the initial response to treatment and identify nonresponders and at 12 weeks is required to see the final response and thus decide upon continuation or discontinuation of treatment. In the follow-up visit at 4 and 12 weeks, CBC, Iron profile (Iron, Ferritin, and TIBC), CRP, and AGP will be done. Corrected Reticulocyte will be done at 4 weeks only. Any adverse effects of therapy will be noted. Adherence to therapy will be checked by measuring the volume of unused medicine in the bottle at each visit. All the statistically analyzed continuous data will be presented as mean ± standard deviation (SD). The categorical data will be reported as a percentage. Student's t-tests will be used to compare means. The χ2 test will be used to compare categorical outcomes, including the proportion of patients with dropouts, adverse effects, and adherence measures. The percentage volume of unused study medication returned at each visit will be compared using the Wilcoxon rank sign test. p<0.05 will be considered statistically significant.

DETAILED DESCRIPTION:
1. Research Hypothesis: Liposomal iron preparation is equally effective and more tolerable than ferrous ascorbate in treating iron deficiency anemia in 6 to 59 months age children.
2. Background & Rationale of the study: Iron deficiency anemia (IDA) is highly prevalent worldwide with underdeveloped and developing countries being most affected. As per the recent NFHS-5 data, 67.1% of 6 to 59 months of age children are anemic in India. About 1/3rd under 5 children reportedly have iron deficiency anemia in India. Poor breastfeeding practices, untimely and improper complementary feeding, predominant milk-based diet, recurrent infections, and low socio-economic status are some of the common risk factors for IDA. Children under 5 years of age are more vulnerable to IDA because of their rapid growth and increased requirement. IDA leads to both short and long-term morbidities including poor appetite, irritability, recurrent infections, and neurodevelopment impairment. Prevention, early diagnosis, and early intervention are keys to managing IDA and thus preventing complications. Ferrous sulphate, ferrous ascorbate, carbonyl iron, polysaccharide iron complex, and liposomal iron are some of the iron preparations which are used as per the personal choice of the treating pediatrician. Poor palatability, untoward gastrointestinal side effects, and staining of teeth are some of the factors which negatively impact compliance with iron therapy. Therefore newer iron preparations need to be explored which can counteract these side effects. Liposomal iron, a form of ferric pyrophosphate is transported within a phospholipid membrane, absorbed by the intestinal M cells, reaches to the liver directly through lymphatics, and is finally released. Due to this mechanism, liposomal iron has been reported to have better bioavailability than traditional iron preparations thus requiring lesser doses and producing fewer adverse effects. Liposomal iron has reportedly been used successfully in the adult population including pregnant females and chronic kidney disease patients. A recent multicentre study has reported that liposomal iron is being used widely in children for IDA. Liposomal iron is given in droplet dispenser form thus facilitating the administration of precise doses in young children. Thus it can be hypothesized that liposomal iron is equally effective as ferrous salts and have better tolerability. However, there is a paucity of studies in the literature on liposomal iron for the treatment of IDA in children. As per our knowledge, there are no randomized controlled trials in the under-5 children group comparing liposomal iron with any other iron preparation. Since ferrous ascorbate is one of the most commonly prescribed iron preparations, therefore this trial would be designed to compare the efficacy of ferrous ascorbate with liposomal iron. The dose of Ferrous ascorbate would be 3mg/kg once daily dosing and the dose of liposomal iron would be 1mg/kg once a day. The dose of drugs was decided as per the WHO recommendations, pediatric textbooks, and recent trials.
3. Preliminary work done if any: No
4. The relevance and the expected outcome of the proposed study: Iron deficiency anemia is highly prevalent in under 5 children in India. Prevention, early diagnosis, and early intervention are the key to managing IDA. Several iron preparations are available across the world. Liposomal iron preparation is expected not to be inferior to commonly used ferrous ascorbate in treating iron deficiency anemia in children. Liposomal iron is also less likely to have common adverse effects associated with other commonly used iron preparations and thus reducing the rate of discontinuation of the medicine.
5. Specific objectives

   Primary objective:

   a. To compare the efficacy of ferrous ascorbate versus liposomal iron for the treatment of nutritional IDA amongst 6 to 59 months age children as determined by the increase in hemoglobin concentration after 12 weeks of treatment

   Secondary objective:
   1. To compare the change in other laboratory parameters of IDA- MCV, corrected reticulocyte count, serum iron, serum ferritin (corrected for markers of inflammation), TIBC, and transferrin saturation between ferrous ascorbate and liposomal iron group.
   2. To compare the adverse effects of drugs between the two groups
   3. To compare the adherence to drugs amongst study subjects in the two groups.
6. Work plan methodology/experimental design to accomplish the stated aim including the sample size (Patient/Control/Volunteers) and source of volunteers/Control:

Study population: children from 6 to 59 months of age attending OPD (outpatient department) of the Pediatrics Department with IDA.

Study design: This study is a randomized, controlled, double-blinded single-center trial to compare the efficacy of ferrous ascorbate versus liposomal iron for the treatment of nutritional IDA in 6 to 59 months age children.

Study setting: outpatient department of Pediatrics of the institute Consent: Written informed consent would be taken from the caregiver

Study protocol:

* Laboratory definition of Anemia: Hemoglobin <11g/dl (as per WHO definition).
* Laboratory definition of IDA:

S No.

Laboratory Tests Performed

Definition of IDA 1. Hemoglobin concentration < 11 gm/dl 2. Mean cell volume (MCV) < 70 µg/dL 3. Serum iron < 30 µg/dL 4a. Serum ferritin (after applying correction factor for CRP and AGP ) ≤ 12 ng/ml 5. Total iron binding capacity (TIBC) > 425 µg/dL 6. Transferrin saturation(Iron×100/TIBC) <16% 7. Corrected reticulocyte count <0.5%

For enrolment in the study patient should have criteria 1& 2 and atleast one of 3,4,5,6

• Correction of Serum Ferritin as per markers of inflammation

Individuals will be categorised into four groups based on their CRP and AGP concentrations:

1. an apparently healthy reference group: (CRP ≤ 5 mg L-1 and AGP ≤ 1gL-1);
2. an incubation group (CRP > 5 mg L-1 and AGP ≤ 1gL-1);
3. an early convalescence group (CRP > 5 mg L-1 and AGP > 1gL-1); and
4. a late convalescence group (CRP ≤ 5 mg L-1 and AGP > 1gL-1). Individual serum ferritin concentrations will then be adjusted by using the relevant, group-specific correction factor(CF) as a multiplier and repeating the calculation . For the incubation group a CF of 0.77 will be used, and for the early and late convalescence groups CFs of 0.53 and 0.75 will be used, respectively.

   * Baseline assessment:

     1. History and physical examination: detailed history including demography, dietary intake of child, any other factors predisposing to IDA, any recent blood transfusion or recent iron therapy, any chronic illness, history of recurrent infections, irritability, poor appetite or any other complication of IDA, history of hypersensitivity to iron would be taken. Complete physical examination including vitals, anthropometry, general and systemic examination would be done.
     2. Laboratory investigations: Complete blood count (CBC), corrected reticulocyte count, Iron Profile (Serum iron, Serum ferritin, serum TIBC) , CRP, AGP and general blood picture.
   * Treatment interventions:

     1. Eligible subjects would be randomized in a 1:1 ratio by computerized software to receive either ferrous ascorbate or liposomal iron.
     2. Subjects in the ferrous ascorbate group would be given drug in dose of 3mg/kg/day OD of elemental iron. Subjects in the liposomal group would be given 1mg/kg/day OD of liposomal iron. In both groups medicine would be given at bedtime. To increase compliance to drug potential negative effects of discontinuing therapy would be clearly explained to the care givers. They would also be told about potential adverse effects of the drug. Strict instructions would be given to caregivers to keep the medicine out of reach of children.
     3. Subjects would be advised to restrict milk intake to less than 500ml and give iron rich foods as per IYCF guidelines.
     4. Follow up visit would be done at 4 and 12 weeks (+2 days). In the follow up visit following points would be noted
   * Any intercurrent illness
   * Any adverse effects of therapy like altered taste, nausea, vomiting, constipation, diarrhea, teeth staining, black stools, abdominal pain
   * Adherence to therapy would be checked by measuring the volume of unused medicine in the bottle at each visit.
   * Dietary history of child will be noted
   * Laboratory studies : CBC, corrected retic count (only at 4 weeks), Iron Profile (serum ferritin, serum iron, TIBC), CRP and AGP.

     5. If at 4 weeks hemoglobin doesn't begin to rise then adherence to drug would be rechecked and re ensured. For such patients repeat hemoglobin will be done at 8 weeks. If hemoglobin rise is <0.5 gm/dl then it would be labeled as treatment failure and that case would be discontinued from study.

     c. Sample size: The sample size calculation is done based on a non-inferiority parallel design. Considering a desired power of 80 %, allocation ratio of 1:1, probability of Type I error of 5 %, common SD for a baseline of 2 g/dl, and the expected clinically relevant difference of 2 g/dl, it was found that a minimum sample of 40 subjects in each arm was sufficient to provide statistically significant results. Considering the dropout rate of 20%, the sample size will be 48 in each group with a total sample size of 96.

     d. Allocation of intervention: randomization of subjects in either group would be done using computerized software in 1:1 ratio. Sequentially numbered opaque sealed envelopes (SNOSE) would be used to effectively conceal the randomization sequence. Subjects and researcher would be blinded to the allocation. Each subject will be given the assigned medicine sufficient for duration of 12 weeks.

     e. Data collection, management and analysis: Clinical information would be collected in the pre tested structured proforma. Details included would be: name, gender, religion, date of birth, current medications, patient's medical and hospitalization history; family history, dietary history, socio economic history, physical examination and laboratory results. Weight and length/height of the subject would be documented. Contact numbers of the primary caregivers will be collected. Amount of unused medicine being brought at each visit will be noted. Data thus collected will be entered in excel sheet. All the statistically analyzed continuous data will be presented as mean ± standard deviation (SD), unless stated otherwise. The categorical data will be reported as a percentage. Student's t tests will be used to compare means. The χ2 test will be used to compare categorical outcomes, including the proportion of patients with dropouts, adverse effects, and adherence measures. The percentage volume of unused study medication returned at each visit will be compared using the Wilcoxon rank sign test. p<0.05 will be considered statistically significant

ELIGIBILITY:
Inclusion Criteria:

Children in the age group 6 to 59 months with Nutritional Iron Deficiency Anaemia as confirmed by hematological parameters

Exclusion Criteria:

1. Subjects with other causes of anemia(hemolytic anemia, bone marrow failure) as evidenced by clinical symptoms and signs and or laboratory values
2. Subjects with ongoing blood loss
3. Subjects who have received any iron therapy or blood transfusion in the past 3 months
4. Subjects with disease interfering with iron absorption e.g. Inflammatory bowel disease, celiac disease, bowel surgery, chronic gastrointestinal infection
5. Subjects with serious chronic medical conditions like chronic kidney disease, congenital heart disease, and chronic lung disease.
6. Subjects with prior history of allergy to iron preparations

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Change in Hemoglobin concentration | 0,4 and 12 weeks
  Change from baseline hemoglobin concentration at 4 and 12 weeks post initiation of therapy

SECONDARY OUTCOMES:
Change in serum ferritin | 0,4 and 12 weeks
  Change from baseline serum ferritin at 4 and 12 weeks post initiation of therapy
Change in Mean corpuscular volume (MCV) | 0,4 and 12 weeks
  Change from baseline MCV at 4 and 12 weeks post initiation of therapy
Change in serum iron | 0,4 and 12 weeks
  Change from baseline serum iron at 4 and 12 weeks post initiation of therapy
Change in total iron binding capacity (TIBC) | 0,4 and 12 weeks
  Change from baseline TIBC at 4 and 12 weeks post initiation of therapy
Change in transferrin saturation | 0,4 and 12 weeks
  Change from baseline transferrin saturation at 4 and 12 weeks post initiation of therapy
Change in corrected reticulocyte count | 0 and 4 weeks
  Change from baseline corrected reticulocyte count at 4 weeks post initiation of therapy
Number of children with adverse effects of drug | 4 and 12 weeks
  Number of children who develop adverse effects of ferrous ascorbate and liposomal iron in respective groups as noted in follow up visits
Volume of unused drug | 4 and 12 weeks
  Adherence to medicine in both groups will be assessed by measuring volume of unused drug brought in follow up visit in each group.

CONTACTS AND LOCATIONS:
Overall Officials: Namita Mishra, MDPediatrics, Principal Investigator — AIIMS Hospital
Locations (1):
- All India Institute of Medical Sciences, Raebareli, Uttar Pradesh, India

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be made available to the journal with whom research will be published
Supporting Information: Study Protocol, SAP
Time Frame: Information will be provided 6 months after data collection is complete and will be available for next 6 months
Access Criteria: Journal with whom research will be published can access the data

REFERENCES:
- [Background] NFHS-5 fact sheets for key indicators based on final data (2019-21) http://rchiips.org/nfhs/NFHS-5_FCTS/India.pdf
- [Background] Sarna A, Porwal A, Ramesh S, Agrawal PK, Acharya R, Johnston R, Khan N, Sachdev HPS, Nair KM, Ramakrishnan L, Abraham R, Deb S, Khera A, Saxena R. Characterisation of the types of anaemia prevalent among children and adolescents aged 1-19 years in India: a population-based study. Lancet Child Adolesc Health. 2020 Jul;4(7):515-525. doi: 10.1016/S2352-4642(20)30094-8. PMID 32562633
- [Background] Mantadakis E, Chatzimichael E, Zikidou P. Iron Deficiency Anemia in Children Residing in High and Low-Income Countries: Risk Factors, Prevention, Diagnosis and Therapy. Mediterr J Hematol Infect Dis. 2020 Jul 1;12(1):e2020041. doi: 10.4084/MJHID.2020.041. eCollection 2020. PMID 32670519
- [Background] Orsango AZ, Habtu W, Lejisa T, Loha E, Lindtjorn B, Engebretsen IMS. Iron deficiency anemia among children aged 2-5 years in southern Ethiopia: a community-based cross-sectional study. PeerJ. 2021 Jun 28;9:e11649. doi: 10.7717/peerj.11649. eCollection 2021. PMID 34249504
- [Background] Zeckanovic A, Kavcic M, Prelog T, Smid A, Jazbec J. Micronized, Microencapsulated Ferric Iron Supplementation in the Form of >Your< Iron Syrup Improves Hemoglobin and Ferritin Levels in Iron-Deficient Children: Double-Blind, Randomized Clinical Study of Efficacy and Safety. Nutrients. 2021 Mar 26;13(4):1087. doi: 10.3390/nu13041087. PMID 33810451
- [Background] Moscheo C, Licciardello M, Samperi P, La Spina M, Di Cataldo A, Russo G. New Insights into Iron Deficiency Anemia in Children: A Practical Review. Metabolites. 2022 Mar 25;12(4):289. doi: 10.3390/metabo12040289. PMID 35448476
- [Background] Guideline: Intermittent Iron Supplementation in Preschool and School-Age Children. Geneva: World Health Organization; 2011. Available from http://www.ncbi.nlm.nih.gov/books/NBK179850/ PMID 24479203
- [Background] Pisani A, Riccio E, Sabbatini M, Andreucci M, Del Rio A, Visciano B. Effect of oral liposomal iron versus intravenous iron for treatment of iron deficiency anaemia in CKD patients: a randomized trial. Nephrol Dial Transplant. 2015 Apr;30(4):645-52. doi: 10.1093/ndt/gfu357. Epub 2014 Nov 13. PMID 25395392
- [Background] Russo G, Guardabasso V, Romano F, Corti P, Samperi P, Condorelli A, Sainati L, Maruzzi M, Facchini E, Fasoli S, Giona F, Caselli D, Pizzato C, Marinoni M, Boscarol G, Bertoni E, Casciana ML, Tucci F, Capolsini I, Notarangelo LD, Giordano P, Ramenghi U, Colombatti R. Monitoring oral iron therapy in children with iron deficiency anemia: an observational, prospective, multicenter study of AIEOP patients (Associazione Italiana Emato-Oncologia Pediatrica). Ann Hematol. 2020 Mar;99(3):413-420. doi: 10.1007/s00277-020-03906-w. Epub 2020 Jan 21. PMID 31965272
- [Background] Bhargava S, Meurer LN, Jamieson B, Hunter-Smith D. Clinical inquiries. What is appropriate management of iron deficiency for young children? J Fam Pract. 2006 Jul;55(7):629-30. PMID 16822452
- [Background] Powers JM, Buchanan GR, Adix L, Zhang S, Gao A, McCavit TL. Effect of Low-Dose Ferrous Sulfate vs Iron Polysaccharide Complex on Hemoglobin Concentration in Young Children With Nutritional Iron-Deficiency Anemia: A Randomized Clinical Trial. JAMA. 2017 Jun 13;317(22):2297-2304. doi: 10.1001/jama.2017.6846. PMID 28609534
- [Background] Ozdemir N. Iron deficiency anemia from diagnosis to treatment in children. Turk Pediatri Ars. 2015 Mar 1;50(1):11-9. doi: 10.5152/tpa.2015.2337. eCollection 2015 Mar. PMID 26078692
- [Background] WHO guideline on use of ferritin concentrations to assess iron status in individuals and populations [Internet]. Geneva: World Health Organization; 2020. Available from http://www.ncbi.nlm.nih.gov/books/NBK569880/ PMID 33909381
- [Background] Nel E, Kruger HS, Baumgartner J, Faber M, Smuts CM. Differential ferritin interpretation methods that adjust for inflammation yield discrepant iron deficiency prevalence. Matern Child Nutr. 2015 Dec;11 Suppl 4(Suppl 4):221-8. doi: 10.1111/mcn.12175. PMID 25721990
- [Background] Visciano B, Nazzaro P, Tarantino G, Taddei A, Del Rio A, Mozzillo GR, Riccio E, Capuano I, Pisani A. [Liposomial iron: a new proposal for the treatment of anaemia in chronic kidney disease]. G Ital Nefrol. 2013 Sep-Oct;30(5):gin/30.5.7. Italian. PMID 24402627
- [Background] Recommendations to prevent and control iron deficiency in the United States. Centers for Disease Control and Prevention. MMWR Recomm Rep. 1998 Apr 3;47(RR-3):1-29. PMID 9563847